CLINICAL TRIAL: NCT06523699
Title: A Pilot Study of the Impact of Recombinant Human Interleukin-7 (CYT107) on Tumor Clearance and Immune Reconstitution in Multiple Myeloma Patients After Autologous Hematopoietic Cell Transplant
Brief Title: Impact of Recombinant Human Interleukin-7 (CYT107) on Tumor Clearance and Immune Reconstitution in Multiple Myeloma Patients After Autologous Hematopoietic Cell Transplant
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Revimmune (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202412127
Record Dates: First submitted 2024-07-22; First posted 2024-07-26 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Multiple Myeloma
Keywords: Myeloma; Immune reconstitution; IL-7; Cytokine; Autologous; Transplant
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Melphalan

STUDY DESIGN:
Intervention Model Description: Randomized 2:1 to receive CYT107 + standard of care melphalan and AHCT or standard of care melphalan and AHCT alone.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- CYT107 + Melphalan + AHCT (Experimental): All patients on this protocol will be treated with standard of care melphalan conditioning followed by autologous hematopoietic stem cell transplant (AHCT). After AHCT, if patients are randomized to the experimental arm, CYT107 will be initiated and will continue for 4 weeks. CYT107 will be administered subcutaneously starting on D+1. Two doses will be given during the first week, and then CYT107 will be administered weekly for 3 more weeks for a total of 5 doses.
  Interventions: Drug: Recombinant glycosylated human interleukin-7; Drug: Melphalan; Procedure: Autologous hematopoietic cell transplant
- Melphalan + AHCT (Active Comparator): All patients on this protocol will be treated with standard of care melphalan conditioning followed by autologous hematopoietic stem cell transplant (AHCT).
  Interventions: Drug: Melphalan; Procedure: Autologous hematopoietic cell transplant

INTERVENTIONS:
Drug: Recombinant glycosylated human interleukin-7 — Provided by RevImmune
  Other Names: CYT107; r-hIL-7
  Arms: CYT107 + Melphalan + AHCT
Drug: Melphalan — Standard of care
Procedure: Autologous hematopoietic cell transplant — Standard of care
  Other Names: AHCT

SUMMARY:
This is a two-arm, open-label, randomized, single-site, pilot study testing the addition of CYT107 following autologous hematopoietic cell transplant (AHCT) in patients with multiple myeloma (MM). The hypothesis of this study is that recombinant human CYT107 can be safely administered after AHCT and will promote quantitative and qualitative T cell reconstitution, which will be associated with enhanced tumor cell clearance and reduced infectious complications. Patients will be randomized to either the intervention arm that will receive CYT107 + standard of care melphalan and AHCT or to the control arm that will receive standard of care melphalan and AHCT only.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of multiple myeloma per IMWG criteria.
* Patient must be in first CR (including CR or sCR) or have PR or VGPR per IMWG criteria.
* Patient must be candidate for melphalan and AHCT in the opinion of the treating physician.
* At least 18 years of age.
* ECOG performance status ≤ 2
* Adequate bone marrow and organ function as defined below:

  * Total bilirubin ≤ 2 x IULN
  * AST(SGOT)/ALT(SGPT) ≤ 2.5 x IULN
  * Creatinine clearance ≥ 30 mL/min by Cockcroft-Gault
* The effects of CYT107 on the developing human fetus are unknown. For this reason and also because many alkylating agents such as melphalan are known to be teratogenic, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for one year post-transplant. Should a woman become pregnant or suspect she is pregnant, or a male suspect he has fathered a child during this time frame, s/he must inform the treating physician immediately.
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* High doses of corticosteroids (greater than 5 mg prednisone equivalent daily) within 2 weeks of Day -2, with exception of premedication as needed for mobilization regimen.
* A history of T-cell malignancy, plasma cell leukemia, or amyloidosis, or history of any other malignancy with the exceptions of in situ carcinomas, non-melanoma skin cancers, and malignancies for which all treatment was completed at least 2 years before Day -2 and the patient has no evidence of disease.
* Currently receiving any other investigational agents.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to CYT107, melphalan, or other agents used in the study.
* Azathioprine, methotrexate, and anti-tumor necrosis factor agents within 2 weeks of Day -2.
* A history of congenital immunodeficiency syndrome or autoimmune disease. Patients with autoimmune disorders adequately controlled with medication (5 mg prednisone equivalent or less) are allowed.
* A history of clinically-significant pulmonary disorders, such as severe asthma, severe COPD, restrictive lung disease, pulmonary embolism within 3 months prior to study enrollment, or active or prior interstitial lung disease/pneumonitis.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative serum or urine pregnancy test within 7 days of Day -2.
* Patients without a backup autologous stem cell graft available.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-04 (Actual); Primary Completion 2029-04-30 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
Rate of non-hematologic grade ≥3 CYT107 treatment-related AEs (excluding expected transplant-related AEs or AEs attributed to melphalan and ASCT) according to CTCAE v5 | Through day 365
  Treatment-related AEs will be defined as AEs occurring that are at least possibly related to the CYT107 treatment, or the combination of melphalan, AHCT, and CYT107.

SECONDARY OUTCOMES:
Rate of minimal residual disease (MRD) | At Day 100
  For the purposes of this study, a patient will be considered as having minimal residual diseases if a positive result (per 10-5 threshold) is obtained using the Adaptive Clonoseq MRD testing.
Rate of response by IMWG of ≥ complete response (CR) | At Day 100
  * Stringent complete response (sCR):
    * CR as defined below
    * Normal free light chain ratio (0.26-1.65)
    * Absence of clonal cells in the bone marrow by immunohistochemistry or immunofluorescence
  * Complete response (CR):
    * Negative immunofixation on the serum and urine
    * <5% plasma cells in the bone marrow aspirate
    * Disappearance of any soft tissue plasmacytomas
Rate of ≥ grade 3 infections | Through day 365
Days from transplant until absolute neutrophil count (ANC) engraftment | Through Day 30
  Neutrophil engraftment is defined as the first day of 3 consecutive days of ANC ≥ 500 following the post-transplant nadir.
Feasibility of treatment schedule | 1 month post-transplant (transplant is on Day 0)
  The study will be feasible if 20% of patients are able to receive all 5 doses of CYT107 within the first month post-transplant.
Absolute lymphocyte count (ALC) recovery from pre-AHCT | Through Day 30

CONTACTS AND LOCATIONS:
Overall Officials: Dilan A Patel, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu